CLINICAL TRIAL: NCT03462966
Title: Effects of Rifaximin on Visceral Hypersensitivity in Irritable Bowel Syndrome
Brief Title: Rifaximin on Visceral Hypersensitivity
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: recruitment challenges
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Principal Investigator, Nipaporn Pichetshote, Staff Physician, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 49509
Record Dates: First submitted 2017-11-20; First posted 2018-03-13 (Actual); Results first posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-08

CONDITIONS: Visceral Hypersensitivity; Irritable Bowel Syndrome
Keywords: Rifaximin; Xifaxan
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Therapeutic (Experimental): 40 subjects with diarrhea-predominant IBS (IBS-D) or mixed IBS (IBS-M) will be enrolled in the study. At the first clinic visit, subjects will undergo rectal sensitivity testing, as well as lactulose breath testing. Subjects will be asked to record their symptoms and bowel habits in a diary over the next 7 days. During the second clinic visit, subjects will receive a 14-day course of rifaximin (550 mg PO TID). During these 14 days, subjects will record their symptoms and bowel habits. Subjects will return to the clinic after completion of the medication and will undergo repeat evaluation via rectal sensitivity testing to assess for change in rectal sensitivity.
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: Rifaximin — Rifaximin will be administered to patients diagnosed with IBS-D or IBS-M to evaluate whether the medication is effective in decreasing rectal hypersensitivity. The secondary objective of the study is to assess the role of SIBO in rectal sensitivity.
  Other Names: Xifaxan

SUMMARY:
Irritable bowel syndrome (IBS) is one of the most common gastrointestinal disorders, with a global prevalence of 11% according to a recent meta-analysis. The total cost of managing IBS in the United States is in excess of $30 billion per year, including indirect costs relating to loss of productivity of more than $20 billion. Abdominal pain/discomfort (i.e. visceral hypersensitivity) is present in all patients with IBS and remains the most therapy-resistant symptom. Apart from abdominal pain, which is measured subjectively using visual scales, several studies have shown a significant increase in rectal sensitivity, which is measured objectively using an inflatable balloon. Drugs which are shown to have objective effects on visceral hypersensitivity are crucial in the management of IBS.

While certain drugs have shown to decrease abdominal pain, there is very little data to substantiate objective changes in visceral hypersensitivity. Rifaximin is a poorly absorbed antibiotic and the exact underlying mechanism of action for rifaximin in reducing the pain component of IBS remains unknown. However, rifaximin has been shown in randomized controlled trials to decrease abdominal discomfort in all subtypes of IBS.

The investigators hypothesize that rifaximin is effective in decreasing rectal visceral hypersensitivity in IBS patients. In this study, the investigators propose to test this hypothesis by measuring visceral hypersensitivity using the graded balloon distention test, before and after a course of rifaximin. To test whether this effect is accompanied by treating SIBO, the investigators will also perform lactulose breath tests before and after rifaximin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18-75 years old inclusive
* Meet Rome IV criteria for IBS-D or IBS-M
* Subjects should report urgency with bowel movement at least once a week
* If subjects are ≥50 years old, a colonoscopy must have been completed within the past 5 years
* Subjects are capable of understanding the requirements of the study, are willing to comply with all the study procedures, and are willing to attend all study visits.
* Agree to use an acceptable method of contraception throughout their participation in the study. Acceptable methods of contraception include: double barrier methods (condom with spermicidal jelly or a diaphragm with spermicide); hormonal methods (e. g. oral contraceptives, patches or medroxyprogesterone acetate); or an intrauterine device (IUD) with a documented failure rate of less than 1% per year. Abstinence or partner(s) with a vasectomy may be considered an acceptable method of contraception at the discretion of the investigator.
* All subjects will provide Institutional Review Board (IRB)-approved informed written consent prior to beginning any study-related activities

NOTE: Female subjects who have been surgically sterilized (e.g. hysterectomy or bilateral tubal ligation) or who are postmenopausal (total cessation of menses for >1 year) will not be considered "females of childbearing potential".

Exclusion Criteria:

* Treatment with antibiotics or Xifaxan in the last two months
* Subjects with history of intestinal surgery (except appendectomy or cholecystectomy)
* Subjects with known pelvic floor dysfunction
* Pregnancy
* Nursing mothers
* Poorly controlled/uncontrolled significant medical condition that would interfere with study procedures
* History of bowel obstruction
* History of celiac disease
* History of inflammatory bowel disease
* Cirrhosis
* IBS-C/chronic idiopathic constipation
* Diabetes
* History of anorectal radiation/surgery
* History of prostatitis
* Known allergy or hypersensitivity to rifaximin or rifamycin
* Current treatment with eluxadoline or opiates

NOTE: Development of any of the exclusion criteria during the study will be considered a basis for subject discontinuation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nipaporn Pichetshote, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Lovell RM, Ford AC. Global prevalence of and risk factors for irritable bowel syndrome: a meta-analysis. Clin Gastroenterol Hepatol. 2012 Jul;10(7):712-721.e4. doi: 10.1016/j.cgh.2012.02.029. Epub 2012 Mar 15. PMID 22426087
- [Background] Cash B, Sullivan S, Barghout V. Total costs of IBS: employer and managed care perspective. Am J Manag Care. 2005 Apr;11(1 Suppl):S7-16. PMID 15926759
- [Background] Low K, Hwang L, Hua J, Zhu A, Morales W, Pimentel M. A combination of rifaximin and neomycin is most effective in treating irritable bowel syndrome patients with methane on lactulose breath test. J Clin Gastroenterol. 2010 Sep;44(8):547-50. doi: 10.1097/MCG.0b013e3181c64c90. PMID 19996983
- [Background] Longstreth GF, Thompson WG, Chey WD, Houghton LA, Mearin F, Spiller RC. Functional bowel disorders. Gastroenterology. 2006 Apr;130(5):1480-91. doi: 10.1053/j.gastro.2005.11.061. PMID 16678561
- [Background] American College of Gastroenterology Task Force on Irritable Bowel Syndrome; Brandt LJ, Chey WD, Foxx-Orenstein AE, Schiller LR, Schoenfeld PS, Spiegel BM, Talley NJ, Quigley EM. An evidence-based position statement on the management of irritable bowel syndrome. Am J Gastroenterol. 2009 Jan;104 Suppl 1:S1-35. doi: 10.1038/ajg.2008.122. No abstract available. PMID 19521341
- [Background] Dalrymple J, Bullock I. Diagnosis and management of irritable bowel syndrome in adults in primary care: summary of NICE guidance. BMJ. 2008 Mar 8;336(7643):556-8. doi: 10.1136/bmj.39484.712616.AD. No abstract available. PMID 18325967
- [Background] Pimentel M, Chow EJ, Lin HC. Eradication of small intestinal bacterial overgrowth reduces symptoms of irritable bowel syndrome. Am J Gastroenterol. 2000 Dec;95(12):3503-6. doi: 10.1111/j.1572-0241.2000.03368.x. PMID 11151884
- [Background] Pimentel M, Chow EJ, Lin HC. Normalization of lactulose breath testing correlates with symptom improvement in irritable bowel syndrome. a double-blind, randomized, placebo-controlled study. Am J Gastroenterol. 2003 Feb;98(2):412-9. doi: 10.1111/j.1572-0241.2003.07234.x. PMID 12591062
- [Background] Lupascu A, Gabrielli M, Lauritano EC, Scarpellini E, Santoliquido A, Cammarota G, Flore R, Tondi P, Pola P, Gasbarrini G, Gasbarrini A. Hydrogen glucose breath test to detect small intestinal bacterial overgrowth: a prevalence case-control study in irritable bowel syndrome. Aliment Pharmacol Ther. 2005 Dec;22(11-12):1157-60. doi: 10.1111/j.1365-2036.2005.02690.x. PMID 16305730
- [Background] Cuoco L, Salvagnini M. Small intestine bacterial overgrowth in irritable bowel syndrome: a retrospective study with rifaximin. Minerva Gastroenterol Dietol. 2006 Mar;52(1):89-95. PMID 16554709
- [Background] Majewski M, McCallum RW. Results of small intestinal bacterial overgrowth testing in irritable bowel syndrome patients: clinical profiles and effects of antibiotic trial. Adv Med Sci. 2007;52:139-42. PMID 18217406
- [Background] Toskes PP. Bacterial overgrowth of the gastrointestinal tract. Adv Intern Med. 1993;38:387-407. No abstract available. PMID 8438647
- [Background] Bouhnik Y, Alain S, Attar A, Flourie B, Raskine L, Sanson-Le Pors MJ, Rambaud JC. Bacterial populations contaminating the upper gut in patients with small intestinal bacterial overgrowth syndrome. Am J Gastroenterol. 1999 May;94(5):1327-31. doi: 10.1111/j.1572-0241.1999.01016.x. PMID 10235214
- [Background] Bures J, Cyrany J, Kohoutova D, Forstl M, Rejchrt S, Kvetina J, Vorisek V, Kopacova M. Small intestinal bacterial overgrowth syndrome. World J Gastroenterol. 2010 Jun 28;16(24):2978-90. doi: 10.3748/wjg.v16.i24.2978. PMID 20572300
- [Background] Posserud I, Stotzer PO, Bjornsson ES, Abrahamsson H, Simren M. Small intestinal bacterial overgrowth in patients with irritable bowel syndrome. Gut. 2007 Jun;56(6):802-8. doi: 10.1136/gut.2006.108712. Epub 2006 Dec 5. PMID 17148502
- [Background] Sachdev AH, Pimentel M. Antibiotics for irritable bowel syndrome: rationale and current evidence. Curr Gastroenterol Rep. 2012 Oct;14(5):439-45. doi: 10.1007/s11894-012-0284-2. PMID 22945316
- [Background] Pimentel M, Lezcano S. Irritable Bowel Syndrome: Bacterial Overgrowth--What's Known and What to Do. Curr Treat Options Gastroenterol. 2007 Aug;10(4):328-37. doi: 10.1007/s11938-007-0076-1. PMID 17761126
- [Background] Pyleris E, Giamarellos-Bourboulis EJ, Tzivras D, Koussoulas V, Barbatzas C, Pimentel M. The prevalence of overgrowth by aerobic bacteria in the small intestine by small bowel culture: relationship with irritable bowel syndrome. Dig Dis Sci. 2012 May;57(5):1321-9. doi: 10.1007/s10620-012-2033-7. Epub 2012 Jan 20. PMID 22262197
- [Background] Nee J, Zakari M, Lembo AJ. Current and emerging drug options in the treatment of diarrhea predominant irritable bowel syndrome. Expert Opin Pharmacother. 2015;16(18):2781-92. doi: 10.1517/14656566.2015.1101449. Epub 2015 Nov 11. PMID 26558923
- [Background] Pimentel M, Chatterjee S, Chow EJ, Park S, Kong Y. Neomycin improves constipation-predominant irritable bowel syndrome in a fashion that is dependent on the presence of methane gas: subanalysis of a double-blind randomized controlled study. Dig Dis Sci. 2006 Aug;51(8):1297-301. doi: 10.1007/s10620-006-9104-6. Epub 2006 Jul 11. PMID 16832617
- [Background] Sharara AI, Aoun E, Abdul-Baki H, Mounzer R, Sidani S, Elhajj I. A randomized double-blind placebo-controlled trial of rifaximin in patients with abdominal bloating and flatulence. Am J Gastroenterol. 2006 Feb;101(2):326-33. doi: 10.1111/j.1572-0241.2006.00458.x. PMID 16454838
- [Background] Pimentel M, Lembo A, Chey WD, Zakko S, Ringel Y, Yu J, Mareya SM, Shaw AL, Bortey E, Forbes WP; TARGET Study Group. Rifaximin therapy for patients with irritable bowel syndrome without constipation. N Engl J Med. 2011 Jan 6;364(1):22-32. doi: 10.1056/NEJMoa1004409. PMID 21208106
- [Background] Pimentel M, Park S, Mirocha J, Kane SV, Kong Y. The effect of a nonabsorbed oral antibiotic (rifaximin) on the symptoms of the irritable bowel syndrome: a randomized trial. Ann Intern Med. 2006 Oct 17;145(8):557-63. doi: 10.7326/0003-4819-145-8-200610170-00004. PMID 17043337
- [Background] Cremonini F, Lembo A. Rifaximin for the treatment of irritable bowel syndrome. Expert Opin Pharmacother. 2012 Feb;13(3):433-40. doi: 10.1517/14656566.2012.651458. Epub 2012 Jan 18. PMID 22251066
- [Background] Di Stefano M, Malservisi S, Veneto G, Ferrieri A, Corazza GR. Rifaximin versus chlortetracycline in the short-term treatment of small intestinal bacterial overgrowth. Aliment Pharmacol Ther. 2000 May;14(5):551-6. doi: 10.1046/j.1365-2036.2000.00751.x. PMID 10792117
- [Background] Mearin F, Lacy BE, Chang L, Chey WD, Lembo AJ, Simren M, Spiller R. Bowel Disorders. Gastroenterology. 2016 Feb 18:S0016-5085(16)00222-5. doi: 10.1053/j.gastro.2016.02.031. Online ahead of print. PMID 27144627
- [Background] Rezaie A, Chua KS, Chang C, et al. Mo2026 Methane on Breath Test Predicts Altered Rectal Sensation During High Resolution Anorectal Manometry. Gastroenterology 2017;146:S-721.
- [Background] van Wanrooij SJ, Wouters MM, Van Oudenhove L, Vanbrabant W, Mondelaers S, Kollmann P, Kreutz F, Schemann M, Boeckxstaens GE. Sensitivity testing in irritable bowel syndrome with rectal capsaicin stimulations: role of TRPV1 upregulation and sensitization in visceral hypersensitivity? Am J Gastroenterol. 2014 Jan;109(1):99-109. doi: 10.1038/ajg.2013.371. Epub 2013 Nov 5. PMID 24189713

RESULTS

PARTICIPANT FLOW:
Recruitment Details: due to recruitment challenges we decided to terminate the clincal trial
Groups:
- Therapeutic: 4 subjects with diarrhea-predominant IBS (IBS-D) or mixed IBS (IBS-M) enrolled in the study. At the first clinic visit, subjects did rectal sensitivity testing, as well as lactulose breath testing. Subjects were asked to record their symptoms and bowel habits in a diary over the next 7 days. During the second clinic visit, subjects will receive a 14-day course of rifaximin (550 mg PO TID). During these 14 days, subjects will record their symptoms and bowel habits. Subjects will return to the clinic after completion of the medication and did repeat evaluation via rectal sensitivity testing to assess for change in rectal sensitivity.
  Rifaximin: Rifaximin will be administered to patients diagnosed with IBS-D or IBS-M to evaluate whether the medication is effective in decreasing rectal hypersensitivity. The secondary objective of the study is to assess the role of SIBO in rectal sensitivity.
Period: Overall Study
Arm/Group | Therapeutic
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Therapeutic
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (14.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4
the mean change in the balloon volume that lead to the first urge to defecate [Mean (Standard Deviation); unit: volume cubic centimeter] | 28 (17.88)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in the Balloon Volume (Measured in Cubic Centimeter) That Leads to First Urge to Defecate.
Description: A 100-cubic centimeter visual analogue scale with verbal descriptors (0=no sensation, 20=first sensation, 40=first sense of urge, 60=normal urge to defecate, 80=severe urge to defecate, and 100=discomfort/pain) will be used to score evoked sensations.
Time Frame: After completing 14-day course of rifaximin.
Measure: Mean (Standard Deviation); unit: volume cubic centimeter
Arm/Group | Therapeutic
Number analyzed (Participants) | 4
volume cubic centimeter | 37.5 (22.17)

2. Secondary Outcome: Association of Urgency Symptom and Rectal Sensitivity Testing.
Description: Association of urgency symptom and rectal sensitivity will be evaluated by the mean change in the balloon pressure (measured in mmHg) that leads to first urge sensation to defecate, evaluated based on the visual analogue scale defined in the primary outcome measure.
Time Frame: After completing 14-day course of rifaximin.
Measure: Mean (Standard Deviation); unit: Millimetre of mercury
Arm/Group | Therapeutic
Number analyzed (Participants) | 4
Millimetre of mercury | 106 (39.29)

3. Secondary Outcome: Number of Participants With a Rise of Hydrogen <20 Parts Per Million Within 90 Minutes of Lactulose Ingestion.(Which is Considered Normal )
Description: Normalization of lactulose breath test as a potential predictor of improvement of rectal hypersensitivity will be evaluated by comparing lactulose breath test results pre- and post-treatment.
  Normalization of lactulose breath test defined as rise of hydrogen <20 Parts per million within 90 minutes of lactulose ingestion.
  patients with positive
Time Frame: After completing 14-day course of rifaximin
Population: Of the 4 participants, only 2 subjects had a breath test post treatment which is needed for this secondary outcome. Both subjects had a normal breath test after treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Therapeutic: Subjects with diarrhea-predominant IBS (IBS-D) or mixed IBS (IBS-M) enrolled in the study(n=4). At the first clinic visit, subjects did rectal sensitivity testing, as well as lactulose breath testing. Subjects were asked to record their symptoms and bowel habits in a diary over the next 7 days. During the second clinic visit, subjects will receive a 14-day course of rifaximin (550 mg PO TID). During these 14 days, subjects will record their symptoms and bowel habits. Subjects will return to the clinic after completion of the medication and did repeat evaluation via rectal sensitivity testing to assess for change in rectal sensitivity.
  Rifaximin: Rifaximin will be administered to patients diagnosed with IBS-D or IBS-M to evaluate whether the medication is effective in decreasing rectal hypersensitivity. The secondary objective of the study is to assess the role of SIBO in rectal sensitivity.
Arm/Group | Therapeutic
Number analyzed (Participants) | 4
Participants | 2

ADVERSE EVENTS:
Time Frame: 1 week and 3 weeks
Arm/Group | Therapeutic
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
recruitment challenges and the COVID pandemic affected our enrollment as we were only able to enroll 4 participants and not all of them finished the outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT03462966/Prot_SAP_001.pdf